CLINICAL TRIAL: NCT05312697
Title: A Phase 2b, Multicenter, Long-term Extension Study of Setrusumab in Adults With Type I, III, or IV Osteogenesis Imperfecta
Brief Title: Long-term Extension Study of Setrusumab in Adults With Type I, III, or IV Osteogenesis Imperfecta
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision not related to safety concerns
Sponsor: Ultragenyx Pharmaceutical Inc (Industry)
Collaborators: Mereo BioPharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: UX143-CL203
Record Dates: First submitted 2022-03-28; First posted 2022-04-05 (Actual); Results first posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Osteogenesis Imperfecta
MeSH Terms: conditions — Osteogenesis Imperfecta | interventions — setrusumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Setrusumab QM -->Setrusumab QM (Experimental): During Retreatment Period: Setrusumab will be administered via intravenous (IV) infusion once a month (QM) for 12 months.
  During Extension Period: Setrusumab will be administered via IV infusion QM for at least 12 months or until commercially available.
  Interventions: Biological: Setrusumab
- Setrusumab QM --> Setrusumab TBD (Experimental): During Retreatment Period: Setrusumab will be administered via IV infusion QM for 12 months.
  During Extension Period: Setrusumab will be administered via IV infusion at a dose frequency to be determined (TBD) for at least 12 months or until commercially available.
  Interventions: Biological: Setrusumab

INTERVENTIONS:
Biological: Setrusumab — A fully human anti-sclerostin monoclonal antibody (mAb)
  Other Names: UX143; BPS804

SUMMARY:
The primary objective of the study is to evaluate bone mineral density (BMD) after 12 months of retreatment with monthly setrusumab in adults with osteogenesis imperfecta (OI).

DETAILED DESCRIPTION:
UX143-CL203 is a long-term extension study in adults with OI who participated in the ASTEROID study (also referred to as MBPS205) [NCT03118570]. The UX143-CL203 study comprises Observation, Retreatment, and Extension Periods. There is no intervention during the Observation Period. During the single-arm Retreatment Period, participants receive open-label setrusumab once a month (QM) for 12 months. Following the Retreatment Period, participants enter an Extension Period in which they will continue treatment with open-label setrusumab at different dosing frequencies.

ELIGIBILITY:
Inclusion Criteria:

* Males or females who participated in the Phase 2b ASTEROID study
* Females of childbearing potential must consent to use highly effective contraception during the Observation, Retreatment, and Extension Periods through 2 months after the last dose of setrusumab and agree not to become pregnant

Exclusion Criteria:

* Known hypersensitivity to setrusumab or its excipients that, in the judgment of the Investigator, places the participant at increased risk for adverse effects
* Presence or history of any condition that, in the view of the Investigator, would interfere with participation, pose undue risk, or would confound interpretation of results
* Pregnant or breastfeeding or planning to become pregnant (self or partner) at any time during the study
* Not willing or able to discontinue bisphosphonates 6 months prior to the Retreatment Screening Visit

Once enrolled in UX143-CL203, individuals who meet any of the following exclusion criteria will not be eligible to participate in the Retreatment Period:

* Concurrent participation in any study that is examining the safety and efficacy of any investigational product or investigational medical device that alters bone health during the Retreatment and Extension Periods, per discretion of the Investigator in consultation with the Medical Monitor.
* Calcium levels outside the normal range at the Retreatment Screening Visit. If the participant's calcium level is not within the normal range, decision to retest should be made in conjunction with the Medical Monitor
* Glomerular filtration rate (GFR) ≤ 29 mL/min at the Retreatment Screening Visit. If the participant's GFR is ≤ 29 mL/min, decision to retest should be made in conjunction with the Medical Monitor
* History of skeletal malignancies or bone metastases at any time
* History of neural foraminal stenosis (except if due to scoliosis)
* History of myocardial infarction, angina pectoris, ischemic stroke or transient ischemic attack (Investigators should consider whether the potential benefits of treatment outweigh the potential risks in patients with other cardiovascular risk factors such as hypertension, hyperlipidemia, familial hyperlipidemia, family history of premature ischemic cardiovascular disease, smoking, diabetes mellitus, and metabolic syndrome.)
* History of or concomitant uncontrolled diseases such as hypo-/hyperparathyroidism, hypo-/hyperthyroidism, Paget's disease, abnormal thyroid function or thyroid disease or other endocrine disorders or conditions that could affect bone metabolism eg, Stage IV/V renal disease
* A history of rickets or osteomalacia or any skeletal condition (other than OI) leading to long-bone deformities and/or increased risk of fractures
* Documented alcohol and/or drug abuse within 12 months prior to dosing or evidence of such abuse as indicated by the laboratory results during the screening/baseline assessments
* Documented history of significant psychiatric or medical disorder that would prevent the participant complying with the requirements of the protocol or would make it unsafe for the participant to participate in the study as judged by the investigator
* Current/previously reported allergy to the study drug or any of its excipients or the class of drug under investigation
* History of external radiation

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2022-04-28 (Actual); Primary Completion 2022-07-07 (Actual); Study Completion 2022-07-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Ultragenyx Pharmaceutical Inc
Locations (1):
- New Mexico Clinical Research & Osteoporosis Center, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Ultragenyx Patient Advocacy/OI Disease Information — https://ultrarareadvocacy.com/conditions-we-study/osteogenesis-imperfecta-oi/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study recruited adults with osteogenesis imperfecta (OI) who previously participated in the phase 2b, double-blind, dose-finding MBPS205 (ASTEROID) study (NCT03118570).
Pre-assignment Details: A total of 2 participants were screened and enrolled. Both participants completed the Baseline visit as part of the Observation Period, and then were discontinued from the study prior to entering the retreatment period as the trial was terminated by the Sponsor.
Groups:
- Observation Period --> Setrusumab QM --> Setrusumab Q2M/Setrusumab Q2M: Following an Observation Period, participants enter a Retreatment Period and receive setrusumab administered via intravenous (IV) infusion once a month (QM) for 12 months. During the planned Extension Period, participants are randomized 1:1 to either continue treatment with open-label setrusumab QM or transition to open-label setrusumab every 2 months (Q2M) for at least 12 months or until setrusumab becomes commercially available.
Period: Overall Study
Arm/Group | Observation Period --> Setrusumab QM --> Setrusumab Q2M/Setrusumab Q2M
Started | 2
Completed | 0
Not Completed | 2
Not completed — Sponsor Terminated Trial | 2

BASELINE CHARACTERISTICS:
Arm/Group | Observation Period --> Setrusumab QM --> Setrusumab Q2M/Setrusumab Q2M
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change From Retreatment Baseline in Lumbar Spine Bone Mineral Density (BMD) Measured by Dual-Energy X-Ray Absorptiometry (DXA) After 12 Months of Setrusumab
Time Frame: Retreatment Baseline, Month 12
Population: No statistical analyses were performed. No primary analysis occurred, as it was planned to occur at the end of the Retreatment Period, reflecting 12 months of retreatment with setrusumab.
Arm/Group | Observation Period --> Setrusumab QM --> Setrusumab Q2M/Setrusumab Q2M
Number analyzed (Participants) | 0

2. Secondary Outcome: Percentage Change From Retreatment Baseline in Total Hip BMD Measured by DXA at Month 12 of the Retreatment Period
Time Frame: Retreatment Baseline, Month 12
Population: as for outcome 1
Arm/Group | Observation Period --> Setrusumab QM --> Setrusumab Q2M/Setrusumab Q2M
Number analyzed (Participants) | 0

3. Secondary Outcome: Annualized New Fracture Rate as Confirmed by Radiograph During the Retreatment Period
Time Frame: Up to Month 12
Population: as for outcome 1
Arm/Group | Observation Period --> Setrusumab QM --> Setrusumab Q2M/Setrusumab Q2M
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From informed consent through early study termination, for an overall mean of 22.5 days
Arm/Group | Observation Period --> Setrusumab QM --> Setrusumab Q2M/Setrusumab Q2M
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is more than 60 days but less than or equal to 180 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-01): https://cdn.clinicaltrials.gov/large-docs/97/NCT05312697/Prot_SAP_000.pdf